CLINICAL TRIAL: NCT02272101
Title: "Rhinitis in the Elderly: A Randomized, Double-Blind, Placebo Controlled, Cross-Over Study of the Effect of Vitamin D Supplementation on Nasal Symptoms and Rhinitis Related Quality of Life"
Brief Title: Rhinitis in the Elderly: The Role of Vitamin D
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rohr and Columbo Asthma, Allergy and Immunology Specialists, P.C. (Other)
Responsible Party: Principal Investigator, Michele Columbo, M.D., Principal Investigator, Rohr and Columbo Asthma, Allergy and Immunology Specialists, P.C.
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: F/N-R14-3326B
Record Dates: First submitted 2013-12-12; First posted 2014-10-22 (Estimated); Last update posted 2014-10-22 (Estimated); Status verified 2014-10

CONDITIONS: Rhinitis
MeSH Terms: conditions — Rhinitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D (Experimental): Vitamin D 4,000 I.U. orally
  Interventions: Dietary Supplement: Vitamin D versus placebo
- Placebo (Placebo Comparator): Placebo orally
  Interventions: Dietary Supplement: Vitamin D versus placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D versus placebo — Cross-over design

SUMMARY:
A study of the role of vitamin D in elderly subjects with perennial and/or nonallergic rhinitis. The hypothesis is that vitamin D supplementation will improve rhinitis symptoms and rhinitis related quality of life.

DETAILED DESCRIPTION:
Rhinitis in the elderly is poorly understood as this group of patients has been ignored in almost all rhinitis studies. Vitamin D deficiency and insufficiency are very common, especially in the elderly. Vitamin D may play an important role in respiratory disease as shown by studies in asthma. This is a randomized, double-blind, placebo controlled, cross-over study. The investigators will look for the effect of vitamin D 4,000 I.U/day vs. placebo for six weeks on symptom scores and rhinitis related quality of life. This study will be performed in the period Nov. 1, 2013 and March 31, 2014, to try to avoid seasonal fluctuations of serum vitamin D due to sun exposure. The investigators will also look for possible associations between serum vitamin D at baseline and study subjects demographics, treatment, and symptom scores.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 65 years old and older with perennial and/or nonallergic rhinitis

Exclusion Criteria:

* Current smokers, digoxin, liver disease, anticoagulants (except for aspirin), planning a surgical procedure during the study period.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Effect of vitamin D on rhinitis symptoms and rhinitis related quality of life measured by standardized questionnaire. | 6 weeks

SECONDARY OUTCOMES:
Associations between baseline serum vitamin D and subjects' demographics and treatment | 6 weeks
  Demographics include age, body mass index, duration of rhinitis, and presence of asthma. Treatment include drugs utilized for treatment of rhinitis expressed as total medication score.

OTHER OUTCOMES:
Safety of vitamin D supplementation in the elderly | 6 weeks
  Will assess serum vitamin D and calcium levels as well as possible side effects from the treatment as reported by the study subjects. No specific tool would be used.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Columbo, M.D., Principal Investigator — Rohr and Columbo Associates
Locations (2):
- United States (2):
  - Rohr and Columbo Asthma, Allergy and Immunology Specialists, P.C., Bryn Mawr, Pennsylvania
  - Rohr and Columbo Asthma, Allergy and Immunology Specialists, Bryn Mawr, Pennsylvania